CLINICAL TRIAL: NCT02440672
Title: A Prospective, Non-randomized, Single Cohort, Multicenter Study to Evaluate the Clinical Outcomes of Total Knee Arthroplasty (TKA) Using the JOURNEY™ II CR Total Knee System
Brief Title: JOURNEY™ II CR Total Knee System
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-4049-06
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; TKA; Degenerative Knee Disease
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Device:JOURNEY™ II CR Total Knee System (J II CR TKS): Subjects having TKA with JOURNEY™ II CR Total Knee System
  Interventions: Device: JOURNEY™ II CR Total Knee System (J II CR TKS)

INTERVENTIONS:
Device: JOURNEY™ II CR Total Knee System (J II CR TKS) — TKA with Journey II CR Total Knee System
  Other Names: JOURNEY™ II CR; (J II CR TKS)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the JOURNEY™ II CR Total Knee System in subjects with degenerative joint disease (DJD) requiring primary total knee replacement.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single cohort, multicenter study to evaluate the clinical outcomes of TKA using the JOURNEY™ II CR Total Knee System in subjects with degenerative joint disease (DJD) requiring primary total knee replacement. One hundred and seventy (170) subjects will be enrolled at up to 18 clinical sites globally. Follow-up clinical assessments will be performed at 3 months, 1 year, 2 years, 5 years, and 10 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST meet ALL of the following criteria for inclusion in the study:

1. Has signed the IRB/EC approved ICF specific to this study prior to study participation
2. Is a male or female ≥ 22 and ≤ 75 years of age presenting with degenerative joint disease (DJD) of the knee
3. Is a candidate for primary total knee arthroplasty with the JOURNEY™ II CR Total Knee System due to DJD, defined by one of the following:

   * Post-traumatic arthritis
   * Osteoarthritis
   * Degenerative arthritis
4. Is able to read and understand the approved Informed Consent Form and Patient Reported Outcome (PRO) assessments (written and oral)
5. Is in general good health (as determined by the Investigator) based on screening assessments and medical history
6. Is independent, ambulatory, and can comply with all post-operative evaluations
7. plans to be available through ten (10) years post-operative follow-up

Exclusion Criteria:

1. Subjects will be excluded from the study, if they meet ANY one (1) of the following criteria:

* Any of the following conditions in the index joint:

  * does not require patella resurfacing
  * has received a TKA or unicondylar arthroplasty
  * has inadequate bone stock to support the device (e.g. severe osteopenia/osteoporosis)
* Any of the following conditions in the contralateral joint:

  * has enrolled in the study for the contralateral knee
  * has received TKA as a revision for a failed total or unicondylar knee arthroplasty
  * has received a primary TKA or unicondylar knee arthroplasty that is not fully healed and well-functioning, as determined by Investigator
  * Any of the following conditions of the hip:
  * received contralateral or ipsilateral revision hip arthroplasty
  * has ipsilateral hip arthritis resulting in flexion contracture
  * has received a ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty, that is not fully healed and well-functioning, as determined by Investigator
  * Has diagnosis of an immunosuppressive disorder
  * Has presence of malignant tumor, metastatic, or neoplastic disease
  * Has family history of severe osteoporosis/osteopenia
  * Has a known allergy to study device or one or more of its components
  * Has conditions that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, lupus, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
  * Is receiving medication for the diagnosis of fibromyalgia
  * has a lower extremity condition causing abnormal or restricted ambulation (e.g. ankle fusion, ankle arthroplasty, previous hip fracture)
  * Is pregnant or plans to become pregnant during the study
  * Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study and complete PROs, as determined by Investigator
  * Has a BMI > 40
  * Is currently enrolled in or has participated in another investigational drug, biologic, or device study within 3 months of enrollment
  * Is currently involved in personal injury litigation or a worker's compensation claim
  * Is facing current or impending incarceration
  * Is known to be at risk for lost to follow-up, or failure to return for scheduled visits

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who present with DJD of the knee will be screened to determine if they meet all inclusion and no exclusion criteria. If all entry criteria are achieved, the subject will be eligible to participate in the study. All general and indication-specific entry criteria must be met prior to study entry.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-09; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Equivalence in 1 year post-operative mean Range of Motion (ROM) in subjects receiving the J II CR TKS as compared to the literature reference mean ROM | 1 year post-op analysis
Non-inferiority of the survival rate of the J II CR TKS with the reference survival rate of a literature reference at 5 and 10-years post-operatively | Up to 10 year post-operative analysis

SECONDARY OUTCOMES:
Clinical Outcomes: EuroQol 5D (EQ-5D) scale | Pre-Op to 10 yrs
Clinical Outcomes: 2011 Knee Society Score (2011 KSS) clinical evaluation | Pre-Op to 10 yrs
Clinical Outcomes: Self-Administered Patient Satisfaction Scale for Primary Hip and Knee Arthroplasty (SAPSS | Pre-Op to 10 yrs
Health Economic Endpoints : Physical therapy visit quantification/duration | 30, 60, and 90-day hospital re-admission rate
Health Economic Endpoints: Discharge destination(s)/length of stay | 30, 60, and 90 days
Health Economic Endpoints: Unscheduled professional visits (e.g. hospital, emergency room, orthopedic clinic, primary care physician) | 30, 60, and 90 days
Health Economic Endpoints: Concomitant medications/procedures associated with the knee | 30, 60, and 90 days
Safety Endpoints:Adverse events, to be evaluated by type, frequency, severity, and relatedness to the study treatment. | Pre-Op to 10 yrs
Safety Endpoints: Manipulations under anesthesia | Pre-Op to 10 yrs
Safety Endpoints: Radiographic analysis | Pre-Op to 10 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Lucy O'Mara, Study Chair — Smith & Nephew, Inc.
Locations (9):
- United States (6):
  - Orthopedic Institute of the West, Phoenix, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - Anne Arundel Health System Research Institute, Inc, Annapolis, Maryland
  - Center for Hip and Knee Replacement at Columbia University Medical Center, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - The Lindner Research Center, Musculo-Skeletal Division - The Christ Hospital Health Network, Cincinnati, Ohio
- Hospital Parc Taulí Servei de Cirurgia Ortopèdica I Traumatologia, Barcelona, Spain
- United Kingdom (2):
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore
  - Barts Health NHS Trust, Whitechapel